CLINICAL TRIAL: NCT06396533
Title: Increasing Pre-Surgical Identification of Muscle Invasive Tumor Evaluations Prior to Planned Cystectomy
Brief Title: Increasing Pre-Surgical Identification of Muscle Invasive Tumor Evaluations Prior to Planned Cystectomy (INSITE)
Acronym: INSITE
Status: Recruiting | Type: Observational
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: GU-222, 24-4001
Record Dates: First submitted 2024-03-27; First posted 2024-05-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Urothelial Carcinoma; Muscle Invasive Bladder Urothelial Carcinoma; Non-Muscle Invasive Bladder Urothelial Carcinoma
Keywords: cystectomy
MeSH Terms: conditions — Carcinoma, Transitional Cell

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urinary genomic biomarker (ctDNA and cfDNA)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non- neoadjuvant chemotherapy patients: Archival (FFPE) specimen of prior diagnostic TUR will be obtained.
  For patients receiving neoadjuvant chemotherapy: Blood will be collected at pre-treatment/baseline, mid-treatment(C3D1), day of cystectomy, and then only serum/plasma 4-6 weeks (±2 weeks) post-cystectomy, and 6 months (±1 month) post-cystectomy.
  For patients not receiving neoadjuvant chemotherapy: Freshly voided mid-stream urine will be collected on the day of cystectomy.
- Neoadjuvant Chemotherapy (NAC) Patients: Archival (FFPE) specimen of prior diagnostic TUR will be obtained.
  For patients not receiving neoadjuvant chemotherapy: Serum/plasma will be collected on the day of cystectomy, and only serum/plasma 4-6 weeks (±2 weeks) post-cystectomy, and 6 months (±1 month) post-cystectomy.
  For patients receiving neoadjuvant chemotherapy: Freshly voided mid-stream urine will be collected from each subject at pre-treatment, mid-treatment (C3D1), and the day of cystectomy.
  Stool samples will be collected in OMNIgene GUT kits. Patients who are not undergoing NAC, will be provided one kit for stool collection prior to cystectomy at baseline. All stool samples will be sent to Case Western Microbiome Core for analysis.

SUMMARY:
This trial aims at investigating the diagnostic ability of a combined diagnostic panel including systematic endoscopic evaluation (SEE), blood-based ctDNA assay, and urine-based cfDNA assay to predict the presence of residual tumor remaining in the bladder at cystectomy.

Patients who are planned for cystectomy due to bladder cancer will be considered for enrollment based on inclusion and exclusion criteria.

DETAILED DESCRIPTION:
The principle outcome of this study is to determine the negative predictive value (NPV) of finding no muscle invasive (pT2) tumor in seeT0 patients with a negative result on the ctDNA assay prior to radical cystectomy.

Eligible candidates for radical cystectomy and INSITE trial:

* Patients with high grade T1 urothelial carcinoma who elect for "early" /upfront cystectomy
* Patients with non-muscle invasive high grade Ta urothelial carcinoma or carcinoma in situ who have relapsed or are refractory / unresponsive to intravesical therapy and have elected to undergo cystectomy
* cT2-T3 muscle invasive urothelial carcinoma (irrespective of receipt of neo-adjuvant chemotherapy) Prior to cystectomy, tissue (transurethral resection of bladder tumor), urine and blood samples will be obtained at baseline for urine biopsy, ctDNA testing and future correlative studies.

After anesthetic induction for radical cystectomy, the patient will undergo rigid cystoscopy with targeted transurethral resection (TUR) of visible tumor or tumor bed, and two additional random bladder biopsies of normal-appearing bladder mucosa. Urine and blood samples will be obtained day of procedure for utilization for urine biopsy, ctDNA, and future correlative studies.

Following cystectomy, a diagnostic testing panel of pre-cystectomy cystoscopic and biopsy findings, ctDNA, and urine biopsy will be compared to final pathologic specimen.

Blood samples will be obtained 4-6 weeks (±2 weeks) post-procedure and 6 months (±1 month) post-procedure for analysis and ctDNA for post-procedure surveillance and other additional correlative studies. Additional blood sample collections at 12 months and 24 months post-procedure are optional.

ELIGIBILITY:
Inclusion Criteria:

1. Properly counselled patients with high grade T1 disease who elect for cystectomy
2. Properly counselled patients with non-muscle invasive high grade Ta urothelial carcinoma or carcinoma in situ who are unresponsive to intravesical therapy and have elected cystectomy
3. cT2-T3 muscle invasive urothelial carcinoma for planned cystectomy
4. Patient who have received prior intravesical therapy or multiple TURBTs can be enrolled (data regarding number of previous TURBTs and type of intravesical therapy will be collected).
5. Male or female patients age >=18 years at the time of consent.
6. Able and willing to comply with study requirements.
7. Patients must have a non-contrast phase component for CT scans of chest/abdomen/pelvis either pre-existing (prior to accrual) or obtained during the screening process.
8. Patients who undergo neoadjuvant systemic therapy for muscle invasive disease must be enrolled before starting systemic therapy.
9. Ability to understand and willingness to sign a written informed consent and HIPAA authorization document.

Exclusion Criteria:

1. Patients who undergo cystectomy with non-curative intent will be excluded.
2. Patients who have undergone previous definitive pelvic radiation for the purpose of treating bladder malignancy.
3. Patients who are pregnant or nursing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are planned for cystectomy due to bladder cancer will be considered for enrollment based on inclusion and exclusion criteria. Eligible patients will have bio specimen collected in accordance with the trial protocol.
Sampling Method: Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2027-04-23 (Estimated); Study Completion 2029-02-23 (Estimated)

PRIMARY OUTCOMES:
Utility of a proprietary urine and blood biomarker test for muscle-invasive bladder cancer presence | 2 years
  Determine the utility of a novel, proprietary combined blood and urinary genomic biomarker (ctDNA and cfDNA) assay in predicting the presence or absence of a muscle-invasive bladder cancer at cystectomy when no disease is identified on systematic endoscopic evaluation (SEE, aka seeT0).
Utility of a DNA test for muscle-invasive bladder cancer presence | 2 years
  Negative predictive value (NPV) of a negative ctDNA and urine-based cfDNA assay to determine the presence or absence of muscle-invasive bladder cancer (pTmi0) on final cystectomy pathology in patients undergoing radical cystectomy with a pre-surgical seeT0 bladder.

SECONDARY OUTCOMES:
Accuracy of surgical specimen DNA test to predict muscle-invasive disease | 2 years
  Determine the accuracy of a negative blood-based ctDNA assay combined with a urinary genomic cfDNA assay to predict the presence or absence of muscle-invasive disease in cystectomy surgical specimen.
Statistical accuracy evaluation of blood-based ctDNA assay for muscle-invasive bladder cancer presence | 2 years
  Negative predictive value (NPV) of blood-based ctDNA assay to determine the presence or absence of muscle-invasive bladder cancer (pTmi0) on final cystectomy pathology in patients undergoing radical cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kutikov, M.D., Principal Investigator — Fox Chase Cancer Center
Locations (2):
- United States (2):
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania